CLINICAL TRIAL: NCT04793165
Title: Is the Artificial Pancreas, Without Carbohydrate Counting, Efficient and Safe for Ambulatory Patients With Type 1 Diabetes
Brief Title: Is the Artificial Pancreas, Without Carbohydrate Counting, Efficient and Safe in an Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Instituto Tecnológico de Buenos Aires (Other); Universidad Nacional de La Plata (Other); Fundación Nuria/Cellex (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 5302
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes; Autoimmune Diabetes
Keywords: diabetes technology; T1DM; artificial pancreas; closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-hybrid closed-loop system (Experimental): To compare two types of treatments:
  During the first 3 days: Previous or conventional, with CSII plus CGM in open loop.
  During the second 3 day period: AP with CSII plus CGM in a closed-loop system, through the ARG algorithm.
  Interventions: Device: Non-hybrid closed-loop system with ARG algorithm

INTERVENTIONS:
Device: Non-hybrid closed-loop system with ARG algorithm — To assess efficacy and safety of non-Hybrid Closed-loop System, without CHO counting

SUMMARY:
This is a pilot, interventional clinical trial to assess the effectiveness and safety of artificial pancreas (AP) using the ARG algorithm closed-loop system in a monitored 3-day period outpatient study. Once the safety of the device has been validated in the open-loop first 3-day period (continuous subcutaneous insulin infusion (CSII) plus continuous glucose monitoring (CGM)) the investigators will move the study to the second 3-day closed-loop period, without carbohydrate (CHO) counting.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with T1DM at least two years ago and has been using an insulin pump and a CGM for at least 6 months prior to the trial first visit
* Patient is >18 and <65 years
* Patient has HbA1c < 10%
* Woman in premenopausal age agrees to use contraceptive methods
* Woman in premenopausal age has negative B-HCG in the tests performed in the trial
* Patient is trained in CHO counting
* Patient has signed informed consent and has the ability to understand the nature and intent of the study including the ability to comply with study procedures and is willing to keep scheduled visits

Exclusion Criteria:

* Patient has been hospitalized for diabetic ketoacidosis in the last 12 months
* Patient has experienced severe hypoglycemia with loss of consciousness in the last 12 months
* Patient has a history of coronary disease or cardiac failure
* Patient with uncontrolled arterial hypertension
* Patient with a condition that makes the researcher believe that it might increase the chance of hypoglycemia
* Patient has symptoms compatible with active infectious disease
* Patient has Cystic Fibrosis
* Pregnant women, or women with the intention of getting pregnant; women breastfeeding
* Patient has been hospitalized for psychiatric treatment in the last 6 months.
* Patient with a diagnosis of adrenal disease
* Patient has abnormal laboratory values for liver function: transaminase > 2x upper limit normal
* Patient has abnormal laboratory values for renal function: GFR < 60 ml/min/1.73m2
* Patient has active gastroparesis
* Patient is under oncological treatment
* Patient has taken acetaminophen 72 hours previous to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness and safety of AP treatment without CHO counting in an outpatient setting. | 3 days
  Percent of time in each range according to sensor glucose readings

SECONDARY OUTCOMES:
To determine the percentage of time with glycemic levels from 70 to 180 mg/dl (time in range). | 3 days
  Percent of time in the target range of 70-180 mg/dl according to sensor glucose readings
To determine, as a safety parameter, the percentage of time with glycemic levels less than 70 mg/dl. | 3 days
  Percent of time in range of less than 70 mg/dl according to sensor glucose readings

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Grosembacher, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Pena R, Colmegna P, Garelli F, De Battista H, Garcia-Violini D, Moscoso-Vasquez M, Rosales N, Fushimi E, Campos-Nanez E, Breton M, Beruto V, Scibona P, Rodriguez C, Giunta J, Simonovich V, Belloso WH, Chernavvsky D, Grosembacher L. Artificial Pancreas: Clinical Study in Latin America Without Premeal Insulin Boluses. J Diabetes Sci Technol. 2018 Sep;12(5):914-925. doi: 10.1177/1932296818786488. Epub 2018 Jul 12. PMID 29998754
- [Derived] Garelli F, Fushimi E, Rosales N, Arambarri D, Mendoza L, Serafini MC, Moscoso-Vasquez M, Stasi M, Duette P, Garcia-Arabehety J, Giunta JN, De Battista H, Sanchez-Pena R, Grosembacher L. First Outpatient Clinical Trial of a Full Closed-Loop Artificial Pancreas System in South America. J Diabetes Sci Technol. 2023 Jul;17(4):1008-1015. doi: 10.1177/19322968221096162. Epub 2022 May 12. PMID 35549733